CLINICAL TRIAL: NCT04553731
Title: The Effects of mHealth Intervention on Health Empower of Overweight and Obese Women's Body Weight During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Medical College (Other)
Responsible Party: Principal Investigator, Chin-Tsung Shen, the Office of Research and Development, Mackay Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LCF-MOST107
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Overweight and Obese Pregnant Women
MeSH Terms: conditions — Overweight | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The mHealth-based program (Experimental): The experimental group used the mHealth app and Mi Smart Band 5 on managing and preventing excessive GWG among overweight and obese women during pregnancy
  Interventions: Behavioral: empowerment program with mHealth
- The standard antenatal treatments with no mHealth-based elements (No Intervention): controls received standard antenatal treatments with no mHealth-based elements

INTERVENTIONS:
Behavioral: empowerment program with mHealth — empowerment program with mHealth
  Arms: The mHealth-based program

SUMMARY:
evaluate the health empowerment program with mHealth to promote physical activity for overweight and obese pregnant women.

DETAILED DESCRIPTION:
This two-phase study develops an mhealth application (app) based on social-cognitive theory (SCT) and evaluates its effectiveness for overweight and obese women, which can help to prevent excessive GWG by enhancing optimal weight and healthy behavior during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

1. pregnant women--who have had, 8-12 weeks
2. pre-pregnancy body mass index > 25 kg/m2

Exclusion Criteria:

-

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Change in body weight and gestational weight gain from pregnancy to 6 months postpartum | The data were collected before the intervention to childbirth: <16 week gestation, second trimester (24-26 weeks), third trimester (34-36 weeks), 6 months postpartum
  measure body weight and calculated according to the IOM guidelines to know their the total and weekly values of excess or achieve the IOM's guidelines.

SECONDARY OUTCOMES:
Change in physical activity before intervention to childbirth | The data were collected before the intervention to childbirth: <16 week gestation, second trimester (24-26 weeks), third trimester (34-36 weeks); The highest total scores was depend the participants' activities of METs.
  pregnancy physical activity questionnaire (PPAQ) was used to measure women's physical activity during pregnancy.
self-efficacy related weight gain | The data were collected before the intervention to childbirth: <16 week gestation, second trimester (24-26 weeks), third trimester (34-36 weeks); The highest total scores was 125.
  self-efficacy in exercise and diet was used to measure
control infant birthweight | The data were collected at childbirth
  measure infant birthweight

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Fang Lee, PhD, Principal Investigator — Mackay Medical College
Locations (1):
- Department of Nursing, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen HH, Hsiung Y, Lee CF, Huang JP, Chi LK, Weng SS. Effects of an mHealth intervention on maternal and infant outcomes from pregnancy to early postpartum for women with overweight or obesity: A randomized controlled trial. Midwifery. 2024 Nov;138:104143. doi: 10.1016/j.midw.2024.104143. Epub 2024 Aug 11. PMID 39154597
- [Derived] Chen HH, Lee CF, Huang JP, Hsiung Y, Chi LK. Effectiveness of a nurse-led mHealth app to prevent excessive gestational weight gain among overweight and obese women: A randomized controlled trial. J Nurs Scholarsh. 2023 Jan;55(1):304-318. doi: 10.1111/jnu.12813. Epub 2022 Sep 19. PMID 36121127